CLINICAL TRIAL: NCT02896829
Title: Follow-up of the Persistence of the Complete Molecular Remission After Stopping Imatinib Chronic Myeloid Leukemia
Acronym: STIM-FU
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2012/06
Record Dates: First submitted 2016-08-17; First posted 2016-09-12 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Imatinib treatment ending: Interruption of the treatment by Imatinib
  Interventions: Behavioral: Interruption of the treatment by Imatinib

INTERVENTIONS:
Behavioral: Interruption of the treatment by Imatinib

SUMMARY:
It's an observational study based on 98 patients included in the STIM trial to extend the monitoring of patients and to have molecular and clinical data, with long follow up. Are there late relapses? What has become patients who relapsed during STIM trial and restarted TKI (inhibitor tyrosine kinase) treatment?

DETAILED DESCRIPTION:
Chronic myeloid leukemia (CML) is an hematopoietic stem cell disorder in which a t (9;22) (q34;q11) reciprocal chromosomal translocation gives rise to Philadelphia chromosome (Ph) and generates the BCR-ABL1 fusion gene encoding a constitutively activated protein tyrosine kinases (PTK). Tyrosine kinase Inibitors (TKIs) such as imatinib, by blocking BCR-ABL1 kinase activity, selectively eradicate CML cells and induce durable responses and prolong survival.

CML patients treated with TKI are monitored by BCR-ABL1 RT-qPCR (Reverse Transcription real-time quantitative Polymerase Chain Reaction) performed from peripheral blood samples.

A first multicenter study entitled STIM trial demonstrated that imatinib could be safely discontinued in patients with complete molecular remission (CMR) for at least 2 years (undetectable BCR-ABL1 transcript by RT-qPCR).

Around 40% of these patients remain in a prolonged treatment-free remission (TFR) after treatment cessation. All molecular relapsing patients were sensitive when imatinib was re-challenged.

The purpose of this STIM-FU study is to follow all the patients included in the STIM trial in order to evaluate their molecular status, vital status and ongoing treatment in patient with a first molecular relapse.

This long term follow up will allow us to predict if a constant long term control of the disease is possible and to better define the clinical and biological CML-related factors predictive for a molecular relapse after TKI discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* The patients should have been included in the STIM1 Study CHUBX 2006/06 (NCT00478985)

Exclusion Criteria:

* The patients not included or discharged prematurely from the STIM1 Study can not participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the STIM1 protocol with persistence of the Complete Molecular Remission after Stopping Imatinib Chronic Myeloid Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2013-04-03 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Assessment of the molecular status (BCR-ABL1 quantification by RT-qPCR) in the STIM1 population who stopped or restart a treatment by tyrosine kinase inhibitor (TKI) | up to five years

SECONDARY OUTCOMES:
Evaluation of rate of molecular relapse after imatinib discontinuation | up to five years
Evaluation of duration of deep molecular response after stopping imatinib | up to five years
Status dead or alive for each patient | up to five years

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHU d'Angers, Angers
  - Institut Bergonié, Bordeaux
  - CHU de Bordeaux - Haut-Lévêque, Bordeaux
  - Hôpital Morvan, Brest
  - Hôpital Henri-Mondor, Créteil
  - Pôle de cancérologie, Grenoble
  - Centre Hospitalier de La Roche Sur Yon, La Roche-sur-Yon
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital Claude Huriez, Lille
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU Hôtel-Dieu, Nantes
  - CHU de Nice, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital Civil, Strasbourg
  - Hôpital Purpan, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No